CLINICAL TRIAL: NCT04705181
Title: The Indications of First Molar Extraction at Tufts University, School of Dental Medicine--A 14-year Retrospective Study
Brief Title: The Indications of First Molar Extraction at Tufts University, School of Dental Medicine
Status: Active, not recruiting | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Bjorn Steffensen, Professor and Chair Department of Periodontology, Tufts University
Other Study IDs: STUDY00000314
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Tooth Extraction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of the present study is to investigate whether there has been a change of criteria for tooth extraction at Tufts University School of Dental Medicine (TUSDM) from 2005 to 2018. The primary outcome is the change of mean of radiographic interproximal bone loss of extracted teeth. The secondary outcomes are changes of other parameters (periodontal, endodontic and restorative) of extracted teeth and reasons for extraction.

DETAILED DESCRIPTION:
The purpose of the present study is to quantitatively evaluate the change in tooth extraction at school setting over the past 14 years.

Aims The aim of the present study is to investigate whether there has been a change of criteria for tooth extraction at Tufts University School of Dental Medicine (TUSDM) from 2005 to 2018. The primary outcome is the change of mean of radiographic interproximal bone loss of extracted teeth. The secondary outcomes are changes of other parameters (periodontal, endodontic and restorative) of extracted teeth and reasons for extraction.

Hypothesis Criteria for extraction of first molar teeth has changed between 2005 and 2018 toward early extraction of teeth with less severe periodontal and other conditions.

Significance Currently, there is not study presenting the quantified data for criteria change for tooth extraction. Also, determining whether to extract a tooth or not actually requires taking several clinical parameters into consideration. The present study will give clinicians a broad review of the change in clinical decision making for tooth extraction.

Materials and Methods Retrospective chart review among patients in TUSDM Pre-doctoral and Post-doctoral Group Practices The study setting is among patients who received dental treatments at TUSDM. The database will be retrospectively reviewed by patients' electronic records in TUSDM Postgraduate (PG) and Undergraduate (UG) clinics from 01/01/2005 till 12/31/2018.

ELIGIBILITY:
Part 1:

Inclusion Criteria:

1. Patients who had fully-erupted first molar extraction (tooth number #3 or #14 or #19 or #30) under Code on Dental Procedures and Nomenclature (CDT) code of D7140 (Extraction, erupted tooth or exposed root) and D7210 (Extraction, erupted tooth requiring removal of bone and/or sectioning of tooth, and including elevation of mucoperiosteal flap if indicated) at TUSDM.
2. The electronic records must include the following data:

   * Gender
   * Age
   * Comprehensive periodontal chart, including probing depth (PD), clinical attachment level (CAL), furcation involvement and mobility. The periodontal chart has to be recorded within 12 months before tooth extraction
   * Periapical radiograph and bite-wing radiographs of extracted tooth. The radiographs have to be taken within 12 months before tooth extraction
   * Reasons for tooth extraction

Part 2:

Inclusion Criteria:

1. Patients who had:

   * Fully-erupted first and second molars (tooth number #2, #3, #14, #15, #18, #19, #30, #31) that were extracted under CDT codes D7140 (Extraction, erupted tooth or exposed root) or D7210 (Extraction, erupted tooth requiring removal of bone and/or sectioning of tooth, and including elevation of mucoperiosteal flap if indicated).
   * The same extracted tooth were replace with dental implant placement under CDT code D6010 (Surgical placement, endosteal implant) within 24 months after extraction.
2. The electronic records must include the following data

   * Sex
   * Age
   * Dental records including:

     * Periapical radiograph of the tooth before extraction: the radiographs have to be taken within 12 months before tooth extraction, including one or more of probing depth (PD), clinical attachment level (CAL), furcation involvement and tooth mobility.

Exclusion Criteria (both parts):

1. Absence of tooth distal to extracted tooth.

   a. Clinical decision for tooth extraction may be affected by tooth location. When the tooth is the distal abutment in the dentition, clinicians tend to keep the tooth even if the prognosis is compromised.
2. Presence of dental implant adjacent to extracted tooth a. Clinical decision for tooth extraction may be affected by adjacent dental implants.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had fully-erupted first molar extraction (tooth number #3 or #14 or #19 or #30) under CDT code of D7140 (Extraction, erupted tooth or exposed root) and D7210 (Extraction, erupted tooth requiring removal of bone and/or sectioning of tooth, and including elevation of mucoperiosteal flap if indicated) at TUSDM
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Change in mean of radiographic interproximal bone loss of extracted teeth | 2005-2018
  * All the measurements are based on the following reference points projected onto the theoretical tooth long axis
    * Cemento-enamel junction (CEJ); if there is dental restoration or prosthesis on tooth making CEJ undetectable on the radiographs, the apical margin of dental restoration or prosthesis will be used as CEJ
    * The most apical points of mesial and distal interproximal bone height
    * The apex of root
  * The radiographic mesial and distal bone loss will be determined by the proportion of the distance between bone height to apex and the distance between CEJ to apex, projected on the tooth axis
  * The greater bone loss of the mesial and distal sides on radiographs will be used for further analysis
Part 2: Change of criteria for tooth extraction | 2007-2018
  The aim for sub-project 2 represent an extension of the Aim for Subproject 1 outlined above. This sub-project will investigate whether there has been a change of criteria for tooth extraction at TUSDM from 2007 to 2018 specifically for and limited to molar teeth that were extracted and subsequently replaced with dental implants.
  Criteria for extraction of first molar teeth has changed between 2007 and 2018 toward early extraction of teeth with less severe periodontal and other conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Steffensen, DDS, MS, PhD, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States